CLINICAL TRIAL: NCT06430502
Title: Clinical Efficacy of Tumour Treatment Vaccine (TTV) Combined With PD-1 in the Treatment of Relapsed Refractory Advanced Solid Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY23189
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Cancer; PD-L1 Gene Mutation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor treatment vaccine combined with PD-1/L1 inhibitor for patients with advanced solid tumors (Experimental): Tumor treatment vaccine(TTV) would be given deep subcutaneously in the arm or near the tumor. Use PD-1/L1 inhibitors in accordance with the drug indication.
  Interventions: Biological: Tumor Treatment Vaccine; PD-1/L1 inhibitors

INTERVENTIONS:
Biological: Tumor Treatment Vaccine; PD-1/L1 inhibitors — Before and after the patient's treatment period using PD-1 inhibitors，patients will receive tumor treatment vaccine(TTV), which would be given deep subcutaneously in the arm or near the tumor.The initial dose is 1ml each time, if the reaction isn't obvious, the dose can be appropriately increased to 2.5-4.0ml each time.The interval between injections can be shortened or extended depending on the patient's condition and response.

SUMMARY:
This study is intended to investigate the clinical efficacy of TTV vaccine combined with PD-1/PD-L1 inhibitor in the treatment of relapsed and refractory advanced solid tumours from a clinical perspective.

DETAILED DESCRIPTION:
The innovative invention of Tumour Treatment Vaccine (TTV) has been verified in previous studies that the TTV vaccine can play a good role in enhancing the anti-tumour effect of immune checkpoint inhibitor therapy, and the tumour suppression rate of combined anti-PD-1 inhibitor reaches 75.96%. Therefore, this study is intended to investigate the clinical efficacy of TTV vaccine combined with PD-1/PD-L1 inhibitor in the treatment of relapsed and refractory advanced solid tumours from a clinical perspective.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years;
2. Subjects must have histologically- or cytologically-confirmed diagnosis of advanced solid tumor(s) and have progressed on or is not eligible for available standard therapy;
3. Subjects have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
4. ECOG score of 0-2, lifespan > 12 weeks;
5. Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
6. Voluntarily participated in this study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. The patient is diagnosed with central nervous system leukemia(symptoms, signs, imaging, cerebrospinal fluid);
2. White blood cell count ≥ 50×10^9/ L or patients with rapid disease progression can't be guaranteed to complete a full treatment cycle;
3. Patients with fungal, bacterial, viral or other uncontrollable infections or requiring four-level isolation treatment.
4. HIV, HBV and HCV positive;
5. Patients with diseases of the central nervous system or autoimmune central nervous system lesions, Including stroke, epilepsy, dementia;
6. Patients have myocardial infection, cardiac angiography or stents, active angina or other obvious clinical symptoms, or have cardiopathic asthma or cardiovascular lymphocytic infiltrates，within 12 months;
7. Patients are on anticoagulation or have severe coagulopathy (APTT>70);
8. Patients in any condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 2weeks prior to investigational drug administration;
9. Patients were infected with covid-19 within 2weeks prior to investigational drug administration;
10. Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator;
11. Subjects in other conditions that are considered unsuitable for this study by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Relief degree of tumors | immediately after the last treatment
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST1.1）

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China